CLINICAL TRIAL: NCT04127058
Title: A Safety/Tolerance Study to Evaluate a New Titration Scheme in Patients With Bipolar I Disorder or Schizophrenia
Brief Title: Evaluating a New Iloperidone Titration Scheme in Bipolar I Disorder or Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VP-VYV-683-1004
Record Dates: First submitted 2019-10-07; First posted 2019-10-15 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Bipolar I Disorder; Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — iloperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CYP2D6 non-poor metabolizers (Other): titrated up to 24 mg daily (12 mg b.i.d.)
  Interventions: Drug: Iloperidone
- CYP2D6 poor metabolizers (Other): titrated up to 12 mg daily (6 mg b.i.d.)
  Interventions: Drug: Iloperidone

INTERVENTIONS:
Drug: Iloperidone — Oral Tablet
  Other Names: FANAPT®; VYV-683

SUMMARY:
This is a single-center open-label study to be conducted in the United States in subjects with bipolar I disorder or schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 to 65 years of age (inclusive)
* Diagnosed with either schizophrenia or bipolar I disorder, manic or mixed type as per DSM-V criteria
* Symptomatically stable within the past two months

Exclusion Criteria:

* Exposure to any investigational medication, including placebo, in the past 60 days
* Non-response to clozapine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2019-11-27 (Actual)

PRIMARY OUTCOMES:
The frequency of treatment-emergent adverse events as measured by the number of events | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Vanda Investigational Site, Marlton, New Jersey, United States